CLINICAL TRIAL: NCT04920487
Title: Prevalence of Gynecological Pathologies and Use of Hormonal Treatments in Women Hospitalized for a Venous Thromboembolic Episode
Acronym: THROMBO-GYN
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: THROMBO-GYN
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of venous thrombosis (venous thromboembolic disease: VTE) in women of childbearing age in France is in the order of 0.3 to 0.5 / 1000 women / year. It is a rare disease, but the majority of events occurring in women of childbearing age are associated with a particular hormonal context (mainly pregnancy and hormonal contraception). VTE is a multifactorial disease and the risk depends on the simultaneous presence of several triggers.

DETAILED DESCRIPTION:
Certain frequent gynecological pathologies are emerging in the literature as new venous thrombotic risk factors independently of hormonal treatment. Indeed, in endometriosis, the prevalence of which is estimated to be around 10%, biological data are in favor of hypercoagulability. Only one epidemiological study has analyzed this parameter. It is a Japanese cohort study in 103,070 pregnant women including 77 VTE during pregnancy. Endometriosis and recurrent pregnancy loss (RPL) were identified as risk factors for VTE (OR: 2.70 (95%CI, 1.21-6.00) for endometriosis and 6.13 (95% 2.48-15.16) for RPL. In polycystic ovary syndrome (PCOS), whose prevalence is estimated at 7-12%, the associated risk of VTE is better known (OR 1.89, 95%CI 1.60-2.24) and was the subject of a recently published meta-analysis in which the principal investigator collaborated. To the investigators knowledge, no study describes the prevalence of gynecological pathologies in women with VTE.

Concerning hormonal contraception, estrogen-progestin contraception (EPC) is widely used in France and is associated with an increase in the risk of VTE of a factor of 3 to 6. After a venous thrombotic episode, EPC is contraindicated, and non-hormonal or progestin-only contraception (POC) can be used. Nevertheless, to date, few studies have focused on the management of hormonal contraceptive treatment at the time of a VTE episode. Moreover, the contraceptive options presented to patients are often based on multiple actors (vascular physicians, gynaecologists, midwives, general practitioners, etc.) and the experience of the VTE episode, for both patients and prescribers, may influence the contraceptive options proposed or chosen, as well as their compliance.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years hospitalized at Saint Joseph Hospital between 01/01/2016 and 12/31/2020 for VTE
* ICD-10 codes I26, I80, I82, O22.3, O22.5.

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this research.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 50 years hospitalized at Saint Joseph Hospital between 01/01/2016 and 12/31/2020 for VTE
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Retrospectively assess the prevalence of gynecological pathologies in women at the time of VTE | Day 1
  Percentage of women with gynecological pathologies at time of VTE

SECONDARY OUTCOMES:
Analyze the characteristics of VTE according to the presence or absence of a gynecological pathology | Day 1
  Characteristics of VTE
Describe of hormone therapy used after VTE | Day 1
  Percentage of women using hormonal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Justine HUGON-RODIN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Mottais-Cosnefroy V, Pecourt M, Yannoutsos A, Fels A, Beaussier H, Alran S, Priollet P, Hugon-Rodin J. Hormone-dependent gynaecological disorders and contraceptive modalities in women with a history of venous thromboembolic event: The THROMBOGYN study. J Med Vasc. 2022 Nov-Dec;47(5-6):228-237. doi: 10.1016/j.jdmv.2022.10.015. Epub 2022 Nov 14. PMID 36464417